CLINICAL TRIAL: NCT06526429
Title: RAPID Local Ischemic Postconditioning in Acute Ischemic Stroke pAtients receiVEd Successful Thrombectomy Reperfusion
Brief Title: Local Ischemic Postconditioning in Acute Ischemic Stroke
Acronym: RAPID-SAVEI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Jiao Tong University Affiliated Sixth People's Hospital (Other)
Collaborators: Zhangzhou Municipal Hospital of Fujian Province (Other); Shanghai East Hospital (Other); RenJi Hospital (Other); First People's Hospital of Hangzhou (Other); Fujian Medical University Union Hospital (Other)
Responsible Party: Principal Investigator, Yueqi Zhu, Professor, Shanghai Jiao Tong University Affiliated Sixth People's Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: RAPID-SAVEI-01-2024
Record Dates: First submitted 2024-07-24; First posted 2024-07-29 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Acute Ischemic Stroke; Mechanical Thrombectomy; Ischemic Postconditioning; Brain Edema; Neuroprotection
MeSH Terms: conditions — Ischemic Stroke; Brain Edema

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Dose 15 (Experimental): Dose 15 involved 5 cycles of blow block and restoration, each for15 seconds.
  Interventions: Procedure: rapid local ischemic postconditioning
- Dose 60 (Experimental): Dose 60 involved 4 cycles of blow block and restoration, each for 60 seconds.
  Interventions: Procedure: rapid local ischemic postconditioning
- Dose 120 (Experimental): Dose 120 involved 4 cycles of blow block and restoration, each for 120 seconds.
  Interventions: Procedure: rapid local ischemic postconditioning
- Dose 180 (Experimental): Dose 180 involved 4 cycles of blow block and restoration, each for 180 seconds.
  Interventions: Procedure: rapid local ischemic postconditioning
- Dose 240 (Experimental): Dose 240 involved 4 cycles of blow block and restoration, each for 240 seconds.
  Interventions: Procedure: rapid local ischemic postconditioning
- Dose 300 (Experimental): Dose 300 involved 4 cycles of blow block and restoration, each for 300 seconds.
  Interventions: Procedure: rapid local ischemic postconditioning

INTERVENTIONS:
Procedure: rapid local ischemic postconditioning — Rapid local ischemic postconditioning (RL-IPostC) is performed immediately (within 5 minutes) after revascularization. A balloon guiding catheter (BGC) positioned on ipsilateral C1 segment of internal carotid artery is inflated and deflated for the temporary occlusion of the antegrade flow.

SUMMARY:
This study aims to determine the safety and optimal dose of rapid local ischemic postconditioning in acute ischemic stroke(AIS) patients received successful thrombectomy reperfusion. In this trial, investigators will halt antegrade cerebral blood flow temporarily by the way of balloon guiding catheter (BGC) inflation/deflation in AIS patients immediately after revascularization. It makes the ischemic reperfusion brain tissue have a capacity of adaptation through intermittent blood flow restoration. The optimal postconditioning intervention dose will be determined for further investigation.

DETAILED DESCRIPTION:
This will be an Bayesian Optimal Interval Phase I/II (BOIN12) trial design to determine the safety and optimal dose of ischemic postconditioning intervention. The BOIN12 design makes the decision of dose escalation and de-escalation by simultaneously taking account of toxicity and efficacy and it quantifies the desirability of a dose in terms of toxicity-efficacy trade off. Under BOIN12, patients are adaptively assigned to the most desirable dose with the optimal toxicity-efficacy trade-off.

Eligible patients are 18 years or older with symptomatic large vessel occluded (LVO) AIS treated with mechanical thrombectomy (MT) achieving successful reperfusion defined as modified thrombolysis in cerebral infarction (mTICI) score 2b or 3. Participants will receive balloon inflation/deflation at ipsilateral C1 segment of internal carotid artery (ICA) for the temporary occlusion of the antegrade blood flow.

Six postconditioning intervention doses were adopted for blocking and restoration of blood blow. This study will include 6 doses with the start dose set at dose 180. Dose 15: 15s/15s, 5 cycles; Dose 60: 60s/60s, 4 cycles; Dose 120: 120s/120s, 4 cycles; Dose 180: 180s/180s, 4 cycles; Dose 240: 240s/240s, 4 cycles; Dose 300: 300s/300s, 4 cycles. In this trial, a maximum number of 60 participants will be enrolled with a cohort size of 5 and cohort number of 12. The maximum sample size of each dose is set at 20.

The safety outcome within 7 days (dose limiting toxicity, DLT) including any one of: 1) malignant middle cerebral artery (MCA) infarction defined as midline shift ≥5 mm at the level of septum pellucidum, or anisocoria attributable to herniation, or death attributable to herniation; 2) procedure related serious adverse events(SAEs); 3) other causally attributable SAEs. Efficacy outcome was patients without clinically meaningful infarction growth at 72 hours (defined as infarction growth<10 mL from baseline to 72 hours).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Presenting with symptoms and signs consistent with acute anterior circulation ischemic stroke
* Pre-stroke modified Rankin Score 0-1
* Baseline National Institute of Health Stroke Scale (NIHSS) score≥6
* Endovascular treatment can be initiated (femoral puncture) within 24 hours from stroke onset (stroke onset time is defined as last known well time)
* Occlusion of the intracranial internal carotid artery, or the middle cerebral artery (MCA) (M1 or M2) and is the culprit artery
* Ischemic core volume is < 70 ml, mismatch ratio is >1.8 and mismatch volume is >15 ml as determined by CT perfusion imaging
* Embolism verified as the etiology of occluded artery and modified Thrombolysis in Cerebral Infarction Score (mTICI) 2b or 3 achieved after mechanical thrombectomy.
* Time from CT perfusion to reperfusion < 2 hours
* Informed consent signed

Exclusion Criteria:

* Stenosis of the proximal middle cerebral artery, internal carotid artery, or common carotid artery (≥50%) of the culprit artery
* Evidence of internal carotid artery lesion that precludes the access and application of balloon guide catheter
* Multiple vascular embolism on different pathways (e.g., bilateral MCA occlusions, or an MCA and a basilar artery occlusion)
* Pre ischemic stroke within past 3 months
* The expected survival time is less than 6 months, could not be followed at 90 days (such as patient with malignant tumor)
* Currently pregnant, mental disease, advanced hepatic and renal insufficiency, severe heart failure
* Participation in other interventional randomized clinical trials that may confound the outcome assessment of the trial
* Other circumstances that the investigator considers inappropriate for this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2024-10-14 (Actual); Primary Completion 2025-07-04 (Actual); Study Completion 2025-07-20 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | within 7 days
  Treatment-Emergent Adverse Events including any one of below:
  1. Malignant middle cerebral artery infarction defined as midline shift ≥5 mm at the level of septum pellucidum, or anisocoria attributable to herniation, or death attributable to herniation.
  2. Complications related to ischemic postcondition intervention that require treatment including distal vascular embolism, local arterial dissection, and local vascular spasm at the intervention site of the internal carotid artery.
  3. Other causally attributable serious adverse events (SAEs)

OTHER OUTCOMES:
Incidence of mitigation on infarction growth | 72 hours after procedure
  Mitigation on infarction growth defined as infarction growth<10 mL from baseline to 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Yueqi Zhu, MD, Principal Investigator — Shanghai Jiao Tong University Affiliated Sixth People's Hospital
Locations (1):
- Shanghai Jiao Tong University Affiliated Sixth People's Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2024-12-23): https://cdn.clinicaltrials.gov/large-docs/29/NCT06526429/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-14): https://cdn.clinicaltrials.gov/large-docs/29/NCT06526429/SAP_001.pdf